CLINICAL TRIAL: NCT00376272
Title: Randomized, Prospective, Parallel Group, Placebo-Controlled, Multi-Center Study on the Use of Valsartan an Angiotensin II AT1-Receptor Blocker in the Prevention of Atrial Fibrillation Recurrence
Brief Title: GISSI-AF - Use of Valsartan an Angiotensin II AT1-Receptor Blocker in the Prevention of Atrial Fibrillation Recurrence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo di Ricerca GISSI (Other)
Responsible Party: Aldo P. Maggioni, Heart Care Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G106
Record Dates: First submitted 2006-09-12; First posted 2006-09-14 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation,atrial remodeling,dysrhythmias,valsartan
MeSH Terms: conditions — Atrial Fibrillation | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Valsartan
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valsartan
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Study purpose The purpose of the study is to show that the addition of valsartan on top of established therapies can reduce the recurrence of atrial fibrillation in patients with a history of recent atrial fibrillation associated with cardiovascular diseases/comorbidities.

Primary objective To demonstrate that, in patients with history of recent atrial fibrillation treated with the best recommended therapies, the addition of valsartan 320 mg is superior to placebo in reducing atrial fibrillation recurrence.

Study design The GISSI-AF is a prospective, multicenter, randomized, double blind, placebo controlled study. Patients with a history of atrial fibrillation will be centrally randomized in a 1:1 ratio to receive either valsartan or placebo.

GISSI-AF will be a pragmatic trial, with broad selection criteria to mimic real clinical practice as much as possible. Since no special examinations or procedures are required for the trial, the economic impact on the National Health Service will be minimized and use of resources likely to be optimized. The enrollment period will last 12 months. The patients will be followed up for 12 months from study entry

All prescribed treatments for AF or for the underlying cardiovascular diseases, including ACE-inhibitors, amiodarone and betablockers, will be allowed:

* patients should be on a stable treatment for at least one month
* the current guideline for hypertension treatment should be applied
* patients should not be started on ARBs during the study

DETAILED DESCRIPTION:
The protocol is sponsored by an independent organization and partially supported by Novartis

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients >=40 years of age
2. Sinus rhythm
3. At least two ECG documented episodes of symptomatic AF in the previous 6 months or After a successful cardioversion for AF performed between 14 days and 48 hours before randomization
4. At least one of the following underlying cardiovascular diseases/comorbidities:

   * heart failure/documented history of LV dysfunction (defined as an EF <40%)
   * history of hypertension >=6 months with/without LVH
   * Type II diabetes mellitus
   * documented history of stroke or peripheral vascular disease
   * documented history of coronary artery disease
   * lone atrial fibrillation with documented LA dilation (LA diameter >=45 mm for men and >=40 mm for women)
5. Written informed consent to participate in the study prior to any study procedures

Exclusion Criteria:

1. Need for a continuous treatment with ARBs for any clinical reasons
2. Contraindications or known hypersensitivity to ARBs
3. Persistent standing systolic blood pressure < 110 mmHg
4. Recent (<6 weeks) acute myocardial infarction or bypass surgery, or percutaneous coronary intervention
5. Clinically significant valvular etiologies
6. Thyroid dysfunction
7. Indication for pacemaker or ICD implant or for an ablative treatment, recent (<6 months) PM or ICD implant, previous ablative treatment
8. Planned cardiac surgery, expected to be performed within 3 months
9. Serum creatinine level above 2.5 mg/dL
10. Significant liver disease
11. Pregnant or lactating women or women of childbearing potential who are not protected from pregnancy by an accepted method of contraception
12. Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety or be associated with poor adherence to the protocol
13. Presence of any non-cardiac disease (e.g. cancer) that is likely to significantly shorten life expectancy
14. Treatment with any investigational agent within 1 month before randomization
15. Currently decompensated heart failure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1442 (Actual)
Dates: Start 2004-11; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To demonstrate that, in patients with history of recent AF treated with the best recommended therapies, the addition of valsartan (titrated up to 320 mg daily) is superior to placebo in reducing over the whole follow-up: | Time to first AF recurrence
First recurrence of AF, | time to first AF recurrence
Rate of patients with more than one AF episode, | end of follow-up

SECONDARY OUTCOMES:
Number of AF episodes | end of fw-up
Number of hospitalizations for CV reasons | end of fw-up
Number of all-cause hospitalizations | end of fw-up
Incidence of thromboembolic events | end of fw-up
Number of patients who die or with non-fatal thromboembolic events | end of fw-up
Number of patients in sinus rhythm at the time of each study visit | end of fw-up
Number of patients in sinus rhythm who did not have any prior AF recurrence during the study | end of fw-up
Duration and characteristics (ventricular rate) of the first recurrence of AF. | end of fw-up

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Disertori, MD, Study Chair — Gruppo di Ricerca GISSI; Roberto Latini, MD, Study Chair — Gruppo di Ricerca GISSI
Locations (113):
- Italy (112):
  - Ospedale Valdichiana Santa Margherita, Cortona, AR
  - Ospedale Cardinal Massaia, Asti, AT
  - Azienda Ospedaliera Giuseppe Moscati, Avellino, AV
  - Ospedale Consorziale Policlinico, Bari, BA
  - Ospedale di Venere, Bari - Carbonara, BA
  - Ospedali Riuniti di Bergamo, Bergamo, BG
  - Ospedale di Bentivoglio, Bentivoglio, BO
  - Ospedale Maggiore, Bologna, BO
  - Ospedale Bellaria, Bologna, BO
  - Casa di Cura Poliambulanza, Brescia, BS
  - Ospedale Civile Mellini, Chiari, BS
  - Ospedlae Generale Regionale, Bolzano, BZ
  - Azienda Ospedaliera G. Brotzu - S. Michele, Cagliari, CA
  - Presidio Ospedaliero Moscati, Aversa, CE
  - Azienda Ospedaliera Sant'Anna e San Sebastiano, Caserta, CE
  - Ospedale Civile Ave Gratia Plena, Piedimonte Matese, CE
  - Ospedale Ave Gratia Plena, San Felice A Cancello, CE
  - Ospedale San Giuseppe e Melorio, Santa Maria Capua Vetere, CE
  - Azienda Ospedaliera Santa Croce e Carle, Cuneo, CN
  - Ospedale Civile Saluzzo, Saluzzo, CN
  - Ospedlae Maggiore, Crema, CR
  - Istituti Ospitalieri di Cremona, Cremona, CR
  - Ospedale Santissima Annunziata, Cosenza, CS
  - Presidio Ospedaliero Mariano Santo, Cosenza, CS
  - Ospedale San Francesco di Paola, Paola, CS
  - Ospedale Santa Barbara, Rogliano, CS
  - Presidio Ospedaliero San Marco Argentano, San Marco Argentano, CS
  - Ospedale Civile "G. Chidichimo", Trebisacce, CS
  - Ospedale Garibaldi - Nesima, Catania, CT
  - Ospedale Civile Pugliese, Catanzaro, CZ
  - Ospedale Civile, Lamezia Terme, CZ
  - Azienda Ospedaliera Mater Domini, Località Germaneto - Catanzaro, CZ
  - Ospedale G. Basilotta, Nicosia, EN
  - Arcispedale Sant'Anna, Ferrara, FE
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli, FI
  - Nuovo Ospedale San Giovanni di Dio, Florence, FI
  - Ospedali Civili di Sampierdarena, Genova-Sampierdarena, GE
  - Ospedale San Carlo, Genova-Voltri, GE
  - Ospedale Civile San Paolo, Monfalcone, GO
  - Ospedale Civile, Imperia, IM
  - Ospedale Civile San Giovanni di Dio, Crotone, KR
  - Presidio Ospedaliero F. Ferrari, Casarano, LE
  - Ospedale Ignazio Veris Delli Ponti, Scorrano, LE
  - Ospedale Civile Bassa Val di Cecina, Cecina, LI
  - Ospedali Riuniti, Livorno, LI
  - Ospedale del dono Svizzero, Formia, LT
  - Ospedale Civile Campo di Marte, Lucca, LU
  - Ospedale Civile, Milazzo, ME
  - Ospedale Carlo Borella, Giussano, MI
  - Ospedale San Raffaele, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Multimedica SPA, Sesto San Giovanni, MI
  - Ospedale Policlinico, Modena, MO
  - Nuovo Ospedale Civile di Sassuolo, Sassuolo, MO
  - Ospedale Madonna delle Grazie, Matera, MT
  - Ospedale Civile, Policoro, MT
  - Ospedale Buccheri La Ferla Fatebenefratelli, Palermo, PA
  - A.R.N.A.S. Ospedale Civico e Benfratelli, Palermo, PA
  - Ospedale V. Cervello, Palermo, PA
  - Presidio Ospedaliero Villa Sofia, Palermo, PA
  - Ospedale Generale Provinciale, Este, PD
  - Ospedale Civile San Massimo, Penne, PE
  - Ospedale Alta Valle del Tevere, Città di Castello, PG
  - Nuovo Ospedale San Giovanni Battista, Foligno, PG
  - Azienda Ospedaliera S. Maria degli Angeli, Pordenone, PN
  - Ospedale Civile, Fidenza, PR
  - Azienda Ospedaliera San Salvatore, Pesaro, PU
  - IRCCS - Fondazione Salvatore Maugeri, Pavia, PV
  - Ospedale Policlinico San Matteo IRCCS, Pavia, PV
  - Csa di Cura Villa Maria Cecilia, Cotignola, RA
  - Ospedale Santa Maria degli Ungheresi, Polistena, RC
  - Policlinico Madonna della Consolazione, Reggio Calabria, RC
  - Ospedale Scillesi D'America, Scilla, RC
  - Ospedali Riuniti Albano-Genzano, Albano Laziale, RM
  - Ospedale San Filippo Neri, Roma, RM
  - CTO, Roma, RM
  - Ospedale San Giovanni, Roma, RM
  - Ospedale San Camillo, Roma, RM
  - Ospedale Sant'Andrea, Roma, RM
  - Ospedale Infermi, Rimini, RN
  - Casa di Cura Madonna della Salute, Porto Viro, RO
  - Presidio Ospedaliero, Rovigo, RO
  - Ospedale G. Fucito, Mercato San Severino, SA
  - Ospedale San Luca, Vallo della Lucania, SA
  - Ospedale San Bartolomeo, Sarzana - Loc. Santa Caterina, SP
  - Ospedale Santa Corona, Pietra Ligure, SV
  - Casa di Cura Villa Verde, Taranto, TA
  - Ospedale SS. Annunziata, Taranto, TA
  - Ospedale Civile G. Mazzini, Teramo, TE
  - Ospedale di Cles, Cles, TN
  - Casa di Cura Villa Bianca, Trento, TN
  - Ospedale Evangelico Valdese, Torino, TO
  - Azienda USL 4 Terni, Terni, TR
  - Ospedale Santa Chiara, Trento, TR
  - Azienda Servizi Sanitari N. 1 Triestina, Trieste, TS
  - Azienda Ospedaliera - Univ. Ospedali Riuniti, Trieste, TS
  - Ospedale De Gironcoli, Conegliano Veneto, TV
  - Ospedale Santa Maria dei Battuti, Conegliano Veneto, TV
  - Ospedale di Ialmicco - Palmanova - Udine, Palmanova, UD
  - Ospedale S. Antonio, San Daniele del Friuli, UD
  - Santa Maria della Misericordia, Udine, UD
  - Azienda Ospedaliera e Universitaria, Varese, VA
  - Ospedale Civile Umberto I, Mestre, VE
  - Ospedale Civile, Mirano, VE
  - Ospedale Civile San Biagio, Bovolone, VR
  - Ospedale G. Fra Castoro, San Bonifacio, VR
  - Presidio Ospedaliero, Soriano Calabro, VV
  - Ospedale Civile G. Jazzolino, Vibo Valentia, VV
  - Ospedale Generale di Zona, Giugliano in Campania
  - Azienda Ospedaliera Vincenzo Monaldi, Napoli
  - Policlinico Universitario Federico II, Napoli
  - Ospedale Santa Maria delle Grazie, Pozzuoli
- Cardiocentro Ticino, Lugano, Switzerland

REFERENCES:
- [Background] Disertori M, Latini R, Maggioni AP, Delise P, Di Pasquale G, Franzosi MG, Staszewsky L, Tognoni G; GISSI-AF Investigators. Rationale and design of the GISSI-Atrial Fibrillation Trial: a randomized, prospective, multicentre study on the use of valsartan, an angiotensin II AT1-receptor blocker, in the prevention of atrial fibrillation recurrence. J Cardiovasc Med (Hagerstown). 2006 Jan;7(1):29-38. doi: 10.2459/01.JCM.0000199778.85343.08. PMID 16645357
- [Background] GISSI-AF Investigators; Disertori M, Latini R, Barlera S, Franzosi MG, Staszewsky L, Maggioni AP, Lucci D, Di Pasquale G, Tognoni G. Valsartan for prevention of recurrent atrial fibrillation. N Engl J Med. 2009 Apr 16;360(16):1606-17. doi: 10.1056/NEJMoa0805710. PMID 19369667
- [Derived] Disertori M, Franzosi MG, Barlera S, Cosmi F, Quintarelli S, Favero C, Cappellini G, Fabbri G, Maggioni AP, Staszewsky L, Moroni LA, Latini R; GISSI-AF investigators. Thromboembolic event rate in paroxysmal and persistent atrial fibrillation: data from the GISSI-AF trial. BMC Cardiovasc Disord. 2013 Apr 15;13:28. doi: 10.1186/1471-2261-13-28. PMID 23586654
- [Derived] Staszewsky L, Wong M, Masson S, Raimondi E, Gramenzi S, Proietti G, Bicego D, Emanuelli C, Pulitano G, Taddei F, Nicolis EB, Correale E, Fabbri G, Bertocchi F, Franzosi MG, Maggioni AP, Tognoni G, Disertori M, Latini R; GISSI-AF Investigators. Left atrial remodeling and response to valsartan in the prevention of recurrent atrial fibrillation: the GISSI-AF echocardiographic substudy. Circ Cardiovasc Imaging. 2011 Nov;4(6):721-8. doi: 10.1161/CIRCIMAGING.111.965954. Epub 2011 Sep 16. PMID 21926261
- [Derived] Disertori M, Lombardi F, Barlera S, Maggioni AP, Favero C, Franzosi MG, Lucci D, Staszewsky L, Fabbri G, Quintarelli S, Bianconi L, Latini R. Clinical characteristics of patients with asymptomatic recurrences of atrial fibrillation in the Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto Miocardico-Atrial Fibrillation (GISSI-AF) trial. Am Heart J. 2011 Aug;162(2):382-9. doi: 10.1016/j.ahj.2011.05.008. Epub 2011 Jul 7. PMID 21835301
- [Derived] Disertori M, Lombardi F, Barlera S, Latini R, Maggioni AP, Zeni P, Di Pasquale G, Cosmi F, Franzosi MG; GISSI-AF Investigators. Clinical predictors of atrial fibrillation recurrence in the Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto Miocardico-Atrial Fibrillation (GISSI-AF) trial. Am Heart J. 2010 May;159(5):857-63. doi: 10.1016/j.ahj.2010.02.016. PMID 20435196
- See also: Related Info — http://www.anmco.it
- See also: Related Info — http://www.gissi.org